CLINICAL TRIAL: NCT06968975
Title: Observational, Real-world, Digital Biomarker, and Integrated Treatment Outcomes in Chronic Inflammatory Demyelinating Polyneuropathy/Polyradiculoneuropathy (CIDP)
Brief Title: Real-world Study of Treatment Outcomes in Chronic Inflammatory Demyelinating Polyneuropathy/Polyradiculoneuropathy (CIDP)
Acronym: ORBIT-CIDP
Status: Recruiting | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS18653
Record Dates: First submitted 2025-04-04; First posted 2025-05-13 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Polyneuropathy, Inflammatory Demyelinating, Chronic
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is an observational, ambispective, descriptive, non-interventional study of people with a chronic inflammatory demyelinating polyneuropathy/polyradiculoneuropathy (CIDP) diagnosis in the United States with residual impairment, disability, or neurological deficits after at least three months of treatment with standard of care therapy. The study is expected to last two years. Enrollment is expected to continue for one year. Depending on when the participant is enrolled, a participant can be followed for between one and two years, through the end of study, approximately two years after the study starts.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

* Neurologist-confirmed diagnosis of CIDP found in the medical record, with the last neurologist visit prior to enrollment containing no information that suggests this diagnosis was reversed
* Active use of at least one of the following CIDP treatments for three months or longer, with no evidence of discontinuation of this therapy as of the last neurologist visit prior to enrollment

  * immunoglobulin
  * corticosteroids, with the exception of prednisone (or equivalent) monotherapy at 10mg or less per day
  * plasma exchange
  * efgartigimod alfa
  * azathioprine
  * mycophenolate mofetil
  * cyclosporine
  * rituximab
  * methotrexate
* Signed informed consent
* Residual impairment, disability, or neurological deficits at enrollment, as defined by a raw I-RODS score of 44 or below

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Evidence of participation in any interventional clinical trial with an investigational drug at the time of enrollment
* Hyperreflexia (increased reflexes) recorded in the medical record during a neurological exam the year before enrollment and after CIDP diagnosis
* Aged under 18 at the time of enrollment

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants living with CIDP with residual disability
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2027-05-17 (Estimated); Study Completion 2027-05-17 (Estimated)

PRIMARY OUTCOMES:
I-RODS score at baseline | Baseline
  The inflammatory Rasch-built overall disability scale (I-RODS) is a 24-item patient-reported questionnaire that captures disease impact on daily tasks with a score ranging from 0 (maximum disability) to 48 (no disability). It contains 24 items across an activity domain and a social participation domain. Each item is rated as "0": Not possible to perform; "1": possible, but with some difficulty, or "2" possible, without any difficulty.
Variations of I-RODS score over the study duration | From Baseline up to End of Study (2 years)
  Difference in I-RODS between baseline and: 6 months after enrollment, 12 months after enrollment, end of study.
  The inflammatory Rasch-built overall disability scale (I-RODS) is a 24-item patient-reported questionnaire that captures disease impact on daily tasks with a score ranging from 0 (maximum disability) to 48 (no disability). It contains 24 items across an activity domain and a social participation domain. Each item is rated as "0": Not possible to perform; "1": possible, but with some difficulty, or "2" possible, without any difficulty.
Variations of I-RODS score after treatment change | From baseline up to End of Study (approx. 2 years)
  Difference in I-RODS tests between the most recent assessments prior to and subsequent to a change in treatment class.
  The inflammatory Rasch-built overall disability scale (I-RODS) is a 24-item patient-reported questionnaire that captures disease impact on daily tasks with a score ranging from 0 (maximum disability) to 48 (no disability). It contains 24 items across an activity domain and a social participation domain. Each item is rated as "0": Not possible to perform; "1": possible, but with some difficulty, or "2" possible, without any difficulty.
Annualized I-RODS response rate | Up to End of Study (approx. 2 years)
  Percent of patients who experienced inflammatory Rasch-built overall disability scale (I-RODS) response over a given time period, normalized to 365 days
Annualized I-RODS relapse rate | Up to End of Study (approx. 2 years)
  Percent of patients who experienced inflammatory Rasch-built overall disability scale (I-RODS) relapse over a given time period, normalized to 365 days

SECONDARY OUTCOMES:
Adjusted INCAT (aINCAT) score at baseline and its variations over the study duration and after treatment change | Baseline and throughout the study (up to 2 years)
  The adjusted score is identical to the inflammatory neuropathy cause and treatment (INCAT) disability score, except for the exclusion of changes in the upper-limb function from 0 (normal) to 1 (minor symptoms or signs in 1 or both arms, but not affecting any of the functions listed in the scale), or from 1 to 0.
Annualized aINCAT response rate | Up to End of Study (approx. 2 years)
  Percent of participants who experienced inflammatory neuropathy cause and treatment (INCAT) response over a given time period, normalized to 365 days
Annualized aINCAT relapse rate | Up to End of Study (approx. 2 years)
  Percent of pparticipantss who experienced inflammatory neuropathy cause and treatment (INCAT) relapse over a given time period, normalized to 365 days
Interobserver variability of remote INCAT assessment | Up to End of Study (approx. 2 years)
  Intraclass correlation coefficient (ICC) will be used to evaluate interobserver variability. ICC value can range from 0 to 1. Values less than 0.5 are indicative of poor reliability, values between 0.5 and 0.75 indicate moderate reliability, values between 0.75 and 0.9 indicate good reliability, and values greater than 0.90 indicate excellent reliability.
Incidence of select comorbidities at baseline and over the study duration | From Baseline up to End of Study (approx. 2 years)
  Number of participants with comorbidity events
Frequency of select comorbidities at baseline and over the study duration | From Baseline up to End of Study (approx. 2 years)
  Events per patient-year
Laboratory measurements at baseline and over study duration | From Baseline up to End of Study (approx. 2 years)
  Complete Blood Count (CBC), serum lipid profile, liver function tests
CAP-PRI score at baseline and its variations over the study duration and after treatment change | From Baseline to End of Study (approx 2 years)
  The chronic acquired polyneuropathy- patient reported index [CAP-PRI(8)] is a participant reported outcome (PRO) that was developed to capture quality of life in people living with neuropathies. It contains 15 items, with a lower score indicating higher quality of life. Each item is rated as "0": not at all; "1": a little bit, or "2" a lot.

CONTACTS AND LOCATIONS:
Locations (1):
- Investigational Site, Swiftwater, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: OBS18653, CIDP Website for potential participants — https://picnichealth.com/care/programs/orbit-cidp